CLINICAL TRIAL: NCT02973425
Title: Take a Break (TAB): mHealth-assisted Skills Building Challenge for Unmotivated Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rajani Sadasivam, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H00007427; R01CA190866-01A1 (NIH); R25CA172009-01A1 (NIH)
Record Dates: First submitted 2016-11-08; First posted 2016-11-25 (Estimated); Results first posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Smoking Cessation
Keywords: mHealth, Smoking cessation,
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NRT and mHealth assessment tool without feedback (Active Comparator): For the comparison group, implementation will be balanced in all variables except the Take a Break Intervention. The investigators will balance the two groups further by having the comparison (NRT-Sampling group) complete mHealth assessments (without feedback or goal-setting) as an attention control.
  Participants randomized to the comparison group will only have access to a mHealth assessment tool similar to the "Challenge Quizzes" but without feedback.
  Interventions: Behavioral: NRT and mHealth assessment tool without feedback
- Take a Break as an augmentation to NRT in Motivation (Experimental): The Intervention: Take a Break as an augmentation to NRT-sampling in Motivation Phase. Take a Break is an intervention in which smokers are encouraged to engage in smoking abstinence. The main element, the "Break," is a two-week challenge where smokers report days they are smoke-free. The Break is preceded by a 1-week training challenge where Challenge Quizzes (ecological momentary assessments) collect information to guide the smokers during the Break. At baseline, all smokers will be provided NRT lozenges for sampling. At weeks 1 and 3 of the "Marathon", our Tobacco Treatment Specialist will call all smokers, assess their experiences and collect data.Participants in the intervention will receive the full tool suite.
  Interventions: Behavioral: Take a Break as an augmentation to NRT-sampling in Motivation Phase

INTERVENTIONS:
Behavioral: Take a Break as an augmentation to NRT-sampling in Motivation Phase — NRT sampling experience & Suite of mHealth motivational tools and mini-games.
  Arms: Take a Break as an augmentation to NRT in Motivation
Behavioral: NRT and mHealth assessment tool without feedback — NRT and mHealth assessment tool without feedback
  Arms: NRT and mHealth assessment tool without feedback

SUMMARY:
Take a Break (TAB) is a randomized trial designed to evaluate Nicotine Replacement Therapy (NRT)-sampling and a mHealth suite of apps. TAB is a time-limited self-efficacy and skills building experience for Motivation Phase smokers. TAB is designed to create a timeline within which motivation smokers will be encouraged to try a brief period of abstinence. Smokers in this Motivation Phase are relatively untapped in research available information. This project offers these smokers point-of-need technology support in the many components of the intervention..

DETAILED DESCRIPTION:
The Take a Break intervention is designed to increase self-efficacy and support new skills for Motivation Phase smokers. We hypothesize that, compared with the NRT-only group, the Take a Break group will have a greater number of days abstinent during the 'break' period, a greater increase in self-efficacy at the end of the 'break' period, a lower time to first quit attempt, and a higher rate of quit at 6 months. This research study will also provide valuable insight into this population of smokers and increase our understanding of which tools may be effective in helping them quit smoking Our Specific Aims are

* AIM 1: Refine the Take a Break mHealth tool and implementation program.
* AIM 2: Conduct a randomized trial of the effectiveness of Take a Break.
* AIM 3: Follow participants in the AIM 2 randomized clinical trial for 6 months to evaluate time to quit attempts, number of quit attempts, and 6-month biochemically verified point prevalent cessation.

ELIGIBILITY:
Inclusion Criteria:

* For all Aims, investigators will include individuals 18 years and older who are identified as current smokers who are not preparing to quit, and are active in care within the UMMHC system, Northwell Health in Long Island, NY, Reliant Medical Group (RMG) in Worcester, MA and Central Western Massachusetts VA (VACWM) in Worcester, MA. Active in care is defined as having at least two clinical visits in the past year. If an eligible participant does not already have a smart phone, one will be provided to them, free of charge, for the duration of their participation in the study.

Exclusion Criteria:

* Exclusion Criteria: Those unwilling to sample nicotine lozenges or participate in the game will be excluded. All patients already on NRT will be excluded. All participants who have a FDA contraindication or cautions for nicotine lozenge use (pregnancy, breastfeeding, recent cardiovascular distress, or phenylketonuria) will be excluded. We have chosen to exclude patients with a diagnosis of depression, due to confounding factors.

Adults unable to consent, individuals who are not yet adults (infants, children, teenagers), and prisoners will be excluded from this study. The Food and Drug Administration (FDA) advises caution for nicotine lozenge use among women who are pregnant. Thus, women who are pregnant at the time of baseline will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajani S Sadasivam, PhD, Principal Investigator — UMMS
Locations (4):
- United States (4):
  - Reliant Medical Group, Worcester, Massachusetts
  - VA Central Western Massachusetts Healthcare System, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Northwell Health, Great Neck, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Houston TK, Chen J, Amante DJ, Blok AC, Nagawa CS, Wijesundara JG, Kamberi A, Allison JJ, Person SD, Flahive J, Morley J, Conigliaro J, Mattocks KM, Garber L, Sadasivam RS. Effect of Technology-Assisted Brief Abstinence Game on Long-term Smoking Cessation in Individuals Not Yet Ready to Quit: A Randomized Clinical Trial. JAMA Intern Med. 2022 Mar 1;182(3):303-312. doi: 10.1001/jamainternmed.2021.7866. PMID 35072714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from UMMHC, Northwell Health, VACWM. Recruitment activities started on November 2016.
Groups:
- NRT and mHealth Assessment Tool Without Feedback: For the comparison group, implementation will be balanced in all variables except the Take a Break Intervention. The investigators will balance the two groups further by having the comparison (NRT-Sampling group) complete mHealth assessments (without feedback or goal-setting) as an attention control.
  Participants randomized to the comparison group will only have access to a mHealth assessment tool similar to the "Challenge Quizzes" but without feedback.
  NRT and mHealth assessment tool without feedback: NRT and mHealth assessment tool without feedback
Period: Overall Study
Arm/Group | NRT and mHealth Assessment Tool Without Feedback | Take a Break as an Augmentation to NRT in Motivation
Started | 220 | 213
Completed | 171 | 160
Not Completed | 49 | 53
Not completed — Lost to Follow-up | 49 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NRT and mHealth Assessment Tool Without Feedback | Take a Break as an Augmentation to NRT in Motivation | Total
Number analyzed (Participants) | 220 | 213 | 433
Age, Categorical [Count of Participants; unit: Participants] — Population: The Row population differs from the Overall because some participants didn't report values on some demographic variables.
  Participants
    number analyzed (Participants) | 212 | 201 | 413
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 169 | 163 | 332
    >=65 years | 43 | 38 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 115 | 223
  Male | 112 | 98 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 15 | 43
  Not Hispanic or Latino | 190 | 197 | 387
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 220 | 213 | 433

OUTCOME MEASURES:

1. Primary Outcome: Time to First Quit Attempt
Description: Time to first quit attempt is measured by participant self-report of number of days from baseline to first quit attempt within a 6 month period. At the 6-month follow-up visit, the dates of all quit attempts were assessed using the Timeline Follow-Back Method and used to calculate time to first quit attempt.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NRT and mHealth Assessment Tool Without Feedback | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 171 | 160
days | 0.89 (1.04) | 1.48 (2.29)
Statistical Analysis 1: Comparison: NRT and mHealth Assessment Tool Without Feedback vs Take a Break as an Augmentation to NRT in Motivation; The primary hypothesis was tested through a time-to-event analysis implemented using Cox proportional hazards models; Test type: Other; p = 0.02, Regression, Cox; Cox Proportional Hazard = 1.68, 95% CI 2-sided [1.09 to 2.60]

2. Secondary Outcome: Change in Self-Efficacy at the End of the 6 Months
Description: Self Efficacy is measured by the Self-Efficacy Questionnaire (SEQ-12).The SEQ-12 is a 12-item instrument (two six-item subscales) that measures the confidence in ability to refrain from smoking when facing internal stimuli (e.g. feeling depressed) and external stimuli (e.g. being with smokers).
  The scale varies from 1-5 [Not at all (1) Not very(2) Moderately(3) Very (4) Extremely (5)] A higher score indicates a higher level of confidence to refrain from smoking in certain social or emotional situations and a lower score indicates a lower level of confidence to refrain from smoking.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: SEQ-12 overall score (mean)
Arm/Group | NRT and mHealth Assessment Tool Without Feedback | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 171 | 160
SEQ-12 overall score (mean) | 2.7 (0.9) | 2.9 (1.0)
Statistical Analysis 1: Comparison: Take a Break as an Augmentation to NRT in Motivation; For hypothesis 3, we compared the mean score on the SEQ-12 and its subscales at 6 months, adjusting for baseline; Test type: Other; p = 0.03, Regression, Linear; Linear regression = 0.03

3. Secondary Outcome: Point Prevalent Cessation as Measured by Carbon Monoxide Levels
Description: Point prevalent cessation here is measured by the number of participants with a decreased carbon monoxide level as verified by carbon monoxide levels in blood.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | NRT and mHealth Assessment Tool Without Feedback | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 171 | 160
Participants | 17 | 28
Statistical Analysis 1: Comparison: NRT and mHealth Assessment Tool Without Feedback vs Take a Break as an Augmentation to NRT in Motivation; Test type: Other — Six-month OR, 95%CI, and P value were calculated from generalized estimating equation marginal models with a logit link and an exchangeable correlation matrix; p = 0.048, Chi-squared — Analysis models were adjusted by study site, having quit attempts in the past 12 months measured at baseline, cigarettes per day measured at baseline, quit attempts in the past 12 months measured at baseline; Odds Ratio (OR) = 1.92, 95% CI 2-sided [1.01 to 3.68]

4. Secondary Outcome: Mean Number of Days Abstinent During the First 3 Weeks
Description: Measure the mean number of days abstinent as self-reported by participant via the mHealth assessment.
Time Frame: 3 Weeks
Population: The number of participants analyzed is higher than the number of participants who completed the study as all participants were able to self-reported the number of days abstinent at three weeks.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NRT and mHealth Assessment Tool Without Feedback | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 209 | 200
days | 0.60 (2.38) | 1.20 (3.02)
Statistical Analysis 1: Comparison: NRT and mHealth Assessment Tool Without Feedback; During the first 3 weeks from randomization, both the Take a Break and comparison groups reported the number of cigarettes smoked daily (by texting); texting response rate (responded on at least 1 day); Test type: Other; p = 0.01, Regression, Linear; Odds Ratio (OR) = 2.01

5. Secondary Outcome: Number of Participants Abstinent During the First 3 Weeks
Description: Number of participants abstinent within the 3 week period as self-reported by participant via the mHealth assessment.
  .
Time Frame: 3 Weeks
Population: The population analyzed includes participants who eventually dropped out.
Measure: Count of Participants; unit: Participants
Arm/Group | NRT and mHealth Assessment Tool Without Feedback | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 209 | 200
Participants | 29 | 49

6. Other Pre Specified Outcome: Number of Participants Completing Daily Challenge Quiz
Description: Participants were asked to complete daily challenge quizzes during the first 3 weeks of participation. The challenge quizzes contained daily self-assessment text messages and motivational replies (intervention only)
Time Frame: 3 weeks
Population: The number of participants analyzed is higher than the number of participants who completed the study as all participants were able to complete daily challenge quizzes at baseline and at three weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 213
Participants | 112

7. Other Pre Specified Outcome: Number of Participants Completing a Call With Study Team to Establish a Smoking Abstinence Goal.
Description: Participants in the Intervention group were asked to participate in a goal-setting call to establish a smoking abstinence goal (typically one to two days of abstinence from cigarettes). The outcome measures the number of participants who completed to goal-setting call.
Time Frame: 1 week
Population: The number of participants analyzed is higher than the number of participants who completed the study as more participants were able to complete goal setting at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 213
Participants | 199

8. Other Pre Specified Outcome: Number of Participants Use of Mobile Health Application (mHealth App) to Manage Nicotine Cravings.
Description: TAB participants were encouraged to use mHealth apps that provide relaxation or distraction to help manage smoking cravings. The study team measured the number of participants used mHealth apps to manage nicotine cravings in a 3 week period.
Time Frame: 3 week
Population: The number of participants analyzed varies from number completed to reflect the number of participants still engaged at 3 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 213
Participants | 159

9. Other Pre Specified Outcome: Number of TAB Participants Setting a Brief Abstinence Goal With the TTS (Tobacco Treatment Specialist)
Description: At one week TAB participants were asked to whether they would like to set an abstinence goal for the following 2-week challenge. The outcome measures the number of participants in the TAB group who set a brief abstinence goal
Time Frame: 2 week
Measure: Count of Participants; unit: Participants
Arm/Group | Take a Break as an Augmentation to NRT in Motivation
Number analyzed (Participants) | 213
Participants | 145

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed for each participant through study completion up to six months.
Description: No Adverse Event
Arm/Group | NRT and mHealth Assessment Tool Without Feedback | Take a Break as an Augmentation to NRT in Motivation
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/213
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/213
Other Adverse Events (participants affected / at risk) | 0/220 | 0/213

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT02973425/Prot_SAP_000.pdf